CLINICAL TRIAL: NCT04785105
Title: Natural History of Asymptomatic Superior Mesenteric Arterial Stenosis Depends on Celiac and Inferior Mesenteric Arteries Status.
Brief Title: Natural History of Asymptomatic Superior Mesenteric Arterial Stenosis.
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: SMA_2020
Record Dates: First submitted 2020-06-22; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2020-06

CONDITIONS: Stenosis
Keywords: SMA; Stenosis; Stenosis on scanner
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient with isolated SMA stenosis: patient with isolated SMA stenosis on initial scanner
  Interventions: Other: No intervention
- patient with both SMA stenosis and CA or/and IMA stenosis: patient with both SMA stenosis and CA or/and IMA stenosis on initial scanner
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study was to evaluate asymptomatic superior mesenteric artery (SMA) stenosis prognosis according to the presence of coeliac artery (CA) and/or inferior mesenteric artery (IMA) associated stenosis.

DETAILED DESCRIPTION:
BACKGROUND: The benefit of preventive treatment for SMA stenosis remains uncertain. The latest guidelines remain unclear given the lack of data in the literature.

ELIGIBILITY:
Inclusion Criteria:

* the presence of coeliac artery (CA) and/or inferior mesenteric artery (IMA) associated stenosis.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * patients with isolated >70% SMA stenosis
  * patients with both SMA stenosis and CA or/and IMA >70% stenosis
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Development of mesenteric disease defined as acute mesenteric ischemia or chronic mesenteric ischemia. | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Groupement Hospitalier Est, Bron, France